CLINICAL TRIAL: NCT01728506
Title: An Internet-based Weight Loss and Exercise Intervention for Breast Cancer Survivors: The iWEB Program
Brief Title: An Internet-based Weight Loss and Exercise Intervention for Breast Cancer Survivors
Acronym: iWEB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Kim Dittus, Assistant Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VCC 1109
Record Dates: First submitted 2012-07-24; First posted 2012-11-19 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: breast cancer survivor; Weight loss; Exercise
MeSH Terms: conditions — Breast Neoplasms; Weight Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weight Loss & Exercise (Experimental): Single arm intervention of a 24 week weight loss and exercise intervention.
  Interventions: Behavioral: Weight Loss and Exercise

INTERVENTIONS:
Behavioral: Weight Loss and Exercise — Internet delivered, behaviorally based weight loss and exercise intervention

SUMMARY:
The purpose of this study is to test the effectiveness of a behavioral weight loss and exercise intervention delivered via the internet at different cancer centers in New England. The investigators hypothesize that participants will lose 7% of their body weight. The research is being done because many women who are treated for breast cancer are overweight and treatment for breast cancer is often accompanied by weight gain. Individuals who are overweight may be more likely to have their breast cancer come back. Also women who exercise at least three hours a week seem to have less chance of their cancer coming back. The investigators hope to identify an effective weight loss and exercise intervention for breast cancer survivors that can be easily accessed by many people.

This study is designed to determine the feasibility of conducting a distantly delivered-weight loss and exercise intervention for patients who have been treated for breast cancer at three cancer centers, and to evaluate the efficacy of an Internet-based behavioral weight loss and exercise intervention delivered to overweight/obese breast cancer survivors in three New England locations.

Participants will be recruited from three New England Cancer Centers - the Vermont Cancer Center, Norris Cotton Cancer Center at Dartmouth University and the University of Massachusetts Cancer Center. Participants from each center will undergo baseline assessments that include diet assessment, body measurements (height, weight, etc), a physical activity assessment and be asked to complete a series of questionnaires.

Patients that meet the minimum requirements will be enrolled on the study. They will participate in weekly on-line "chats" about behavioral and diet modifications led by a qualified facilitator. Participants will also engage in increasing amounts of aerobic activity (typically walking) throughout the course of the intervention. The intervention lasts 6 months. At the end of those 6 months, participants will have the same assessments that were collected at baseline. Following the collection of those assessments, participants will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer diagnosis
* Completion of surgery, chemotherapy +/- radiation for stage I, II, or III breast cancer 2-12 months prior to study initiation
* BMI between 27 and 50
* patient self-report of ability to walk for 10 minutes without interruption or pain
* access to computer and the internet

Exclusion Criteria:

* metastatic disease
* prior receipt of chemotherapy for other malignancy
* pregnancy at the time of study entry
* limited food choices due to celiac sprue or inflammatory bowel disease
* illiteracy
* non-English speaking

Ages: 21 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Change from baseline fesability at 6 months
  Feasibility will be determined by length of time required to obtain approval at all three sites, Numbers approached vs. numbers who participate in the study.
Change in diet measures | Change from baseline diet measures at 6 months
  Efficacy will be measured using total calories and fat grams before and after the intervention
Change in anthropometric measures | Change from baseline anthropometrics at 6 months
  Change in Weight, BMI, body fat percentage before and after the intervention
Change in active energy expenditure (ie exercise) | Change from baseline active energy expenditure at 6 months
  exercise will be measured using an accelerometer before and after the intervention

SECONDARY OUTCOMES:
Change in inflammatory biomarkers | Change from baseline inflammatory biomarkers at 6 months
  Change in Il-6, hsCRP before and after the intervention
Change in insulin resistance markers | Change from baseline insulin resistance markers at 6 months
  Change in Homeostatic model assessment to estimate beta cell function and insulin resistance before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Dittus, MD PhD, Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - University of Massachusetts, Worcester, Massachusetts
  - Dartmouth Hitchcock Medical Center, Hannover, New Hampshire
  - Unviersity of Vermont/Fletcher Allen Health Care, Burlington, Vermont